CLINICAL TRIAL: NCT06942195
Title: Effects of Intraduodenal Calcium on Plasma Glucose, Glucoregulatory Hormones and Gastric Emptying in Response to a Mixed-nutrient Drink in Humans With Type 2 Diabetes
Brief Title: Effects of Calcium on Gut Functions and Blood Glucose in Humans With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Christine Feinle-Bisset, Professor Christine Feinle-Bisset, University of Adelaide
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 13243-1
Record Dates: First submitted 2025-04-08; First posted 2025-04-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-04

CONDITIONS: T2DM
Keywords: Intraduodenal; Calcium; Gastric emptying; Glucoregulatory hormones; Plasma glucose; Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In order to blind both investigator and participant, the treatments will be prepared on the morning of each study day, by a research officer who will have no involvement in data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ca-1000 (Active Comparator): In this arm, participants will receive a 75-minute intraduodenal infusion of an isotonic solution containing 3.68 g of calcium chloride dihydrate (CaCl₂·2H₂O), dissolved in 225 mL of distilled water.
  Interventions: Other: Ca-1000
- Ca-500 (Active Comparator): In this arm, participants will receive a 75-minute intraduodenal infusion of an isotonic solution containing 1.84 g of calcium chloride dihydrate (CaCl₂·2H₂O), dissolved in 225 mL of distilled water. Additionally, 1.2 g of sodium chloride (NaCl) will be added to ensure the solution is isosmotic (300 mOsm).
  Interventions: Other: Ca-500
- Control (Placebo Comparator): In this arm, participants will receive a 75-minute intraduodenal infusion of saline (an isotonic solution containing 2.8 g of sodium chloride (NaCl), dissolved in 225 mL of distilled water).
  Interventions: Other: Control

INTERVENTIONS:
Other: Ca-1000 — Calcium, an essential mineral and a key component of dairy, is a regular part of our daily diet. Recent studies have shown that calcium, at doses of 1000 mg, stimulates gut hormones and motility, will be 'higher dose' in this condition.
  Arms: Ca-1000
Other: Ca-500 — Calcium, an essential mineral and a key component of dairy, is a regular part of our daily diet. Recent studies have shown that calcium, at doses of 500 mg, stimulates gut function. In this condition, it will be considered 'lower dose.'
  Arms: Ca-500
Other: Control — Saline (an isotonic solution containing 2.8 g of sodium chloride (NaCl), dissolved in 225 mL of distilled water).
  Arms: Control

SUMMARY:
The intervention in this study consists of a 75-min intraduodenal infusion of an isotonic solution containing either of calcium chloride (CaCl2) or control (saline).

Participants enrolled into the study will receive, in randomised, double-blind fashion (i) Saline (control), (ii) 500 mg CaCl2, or (iii) 1000 mg CaCl2 in three separate sessions, each of which will be separated by at least 4 (and up to 10) days. Each study session will be 4-6 hours. Studies will be carried out in the Clinical Research Facility of the Adelaide Medical School, the University of Adelaide, by staff and students trained in the required techniques.

DETAILED DESCRIPTION:
Each participant will be required to consume a standardised dinner meal (beef lasagne; total energy content: 602 kcal; McCain Food, Wendouree, Victoria, Australia) on the night before each visit by 7 pm. After fasting overnight for ~ 13.5 hours and refraining from exercise and alcohol during the previous 24 hours, the participant will arrive in the laboratory at 8.30 am. After confirming adherence to the study requirements, vital signs ( blood pressure, heart rate and body temperature) will be measured to establish baseline values for safety, and they will be monitored throughout the study. Then, a manometric catheter will be inserted through an anaesthetised nostril and allowed to pass through the stomach and into the duodenum by peristalsis. The infusion port will be positioned ~ 14 cm distal to the pylorus. The correct positioning of the catheter will be monitored continuously by measurement of the transmucosal potential difference in the stomach (~ -40 mV) and the duodenum (~ 0 mV). Once the catheter has been positioned correctly, an intravenous cannula will be placed into a forearm vein for regular blood sampling. At time = -30 minute, a baseline blood sample (7 ml), visual analogue scale (VAS) questionnaire to assess gastrointestinal (GI) symptoms, and breath sample to assess gastric emptying will be collected. Then the infusion of one of the study treatments, i.e. i) saline, ii) 500 mg CaCl2 or iii) 1000 mg CaCl2), will commence and continue for 75 minutes (times = -30 to 45 minutes). At time = -1 minute, participants will consume, within 1 minute, a mixed-nutrient drink (350 mL, containing 500 kcal, 74 g carbohydrates) labelled with 100 mg 13C-acetate for measurement of gastric emptying by non-invasive breath sampling at regular intervals, for subsequent analysis of 13CO2 levels. Blood samples for the measurement of plasma glucose and hormone concentrations, and VAS questionnaires, will be collected before and after the mixed-nutrient drink. At time = 240 minute, after collecting final blood and breath samples and VAS questionnaire, the intravenous cannula will be removed and the participant will be served a light lunch, after which they will be allowed to leave the laboratory. A total of 98 mL of blood (14 sampling time points, 7 mL each) will be taken on each study day (study total of 310 mL, including screening and glucose tolerance test samples).

ELIGIBILITY:
Inclusion Criteria:

* Males with type 2 diabetes mellitus (T2DM). Diagnosis of T2DM will be based on WHO criteria. Only males will be included to avoid the confounding effects of the menstrual cycle on gastric emptying.
* BMI: 28-38 kg/m².
* HbA1c >=6.5 - <=7.9% at screening.
* Blood glucose medications will be required to be withheld for 48 hours prior to each study day.
* Weight-stable (i.e. <5% fluctuation) at study entry, which will be ascertained by a stable body weight in the preceding 3 months.

Exclusion Criteria:

* Significant GI symptoms, or history of GI disease or surgery
* Current gallbladder or pancreatic disease
* Cardiovascular or respiratory diseases
* Any other illnesses (except type 2 diabetes) as assessed by the investigator - (including chronic illnesses not explicitly listed above)
* Use of prescribed or non-prescribed medications (including vitamins and herbal supplements) which may affect energy metabolism, GI function, bodyweight or appetite (e.g. domperidone, cisapride, anticholinergic drugs (e.g. atropine), metoclopramide, erythromycin, hyoscine, orlistat, green tea extracts, Astragalus, St Johns Wort etc.)
* Lactose intolerance/other food allergy(ies)
* Individuals with low ferritin levels (<30 ng/mL), or who have donated blood in the 12 weeks prior to taking part in the study
* High performance athletes
* Current intake of > 2 standard drinks on > 5 days per week (>140g/week)
* Current smokers of tobacco (cigarettes, cigars, pipes, sheesha, chewing, vaping etc.)
* Current use of recreational drugs, e.g. marijuana
* Current intake of any illicit substance
* Vegetarians
* Inability to tolerate nasoduodenal tube
* Inability to comprehend study protocol
* HbA1c <6% or >7.9%
* Estimated glomerular filtration rate <45 ml/min
* Any patient whose medication cannot be withheld for 48 hours for medical reasons

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose concentrations | Blood samples will be collected over 4.5 hours: at baseline (time = -30 minutes), then at regular intervals before and after drink administration (times = -25, -15, 0, 10, 20, 30, 45, 60, 75, 90, 120, 180, 240 minutes).
  Plasma glucose concentrations (mmol/L) will be assessed using glucose oxidase method.

SECONDARY OUTCOMES:
Gastric emptying | Breath samples will be collected in sealed tubes over 4.5 hours: at baseline (time = -30 minutes) (prior to treatment administration), every 5 minutes after the drink (times = 0 to 60 minutes), then every 10 minutes until 240 minutes post-drink.
  13C-acetate breath test, measuring 13CO2 concentrations in end-expiratory breath samples.
Plasma concentrations of glucoregulatory hormones e.g. glucagon-like peptide (GLP-1), glucose-dependent insulinotropic polypeptide (GIP), C-peptide, glucagon, insulin and cholecystokinin (CCK) | Blood samples will be collected over 4.5 hours: at baseline (time = -30 minutes), then at regular intervals before and after the drink (times = -25, -15, 0, 10, 20, 30, 45, 60, 75, 90, 120, 180, 240 minutes).
  Plasma concentration of hormones e.g. GLP-1, GIP and CCK (pmol/L) will be determined using radioimmunoassays, and plasma C-peptide, glucagon and insulin concentrations (pmol/L) will be measured using ELISA immunoassays.
GI symptoms (nausea and bloating) will be assessed as a composite secondary outcome. | Visual Analogue questionnaires will be collected over 4.5 hours: at baseline (time = -30 minutes), at regular intervals before and after the drink (times = -25, -15, 0, 20, 30, 45 minutes), then every 10 minutes until 240 minutes.
  These will be measured using 100mm VAS questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Christine Feinle-Bisset, Principal Investigator — Adelaide Medical School University of Adelaide Level 5 Adelaide Health and Medical Sciences Building, Cnr George St and North Tce, Adelaide, SA 5005
Locations (1):
- Clinical Research Facility, Adelaide Health and Medical Sciences Building, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are not publicly available due to the ethical statement and informed consent that require privacy of data.